CLINICAL TRIAL: NCT05123170
Title: Comparison of Two Different Doses of Dexmedetomidine Added to Lignocaine in Patients Posted for Upper Limb Orthopedic Surgery Under Intravenous Regional Anaesthesia
Brief Title: Dexmedetomidine in IVRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2/2020ANET11
Record Dates: First submitted 2021-10-25; First posted 2021-11-17 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Regional Anesthesia Morbidity
Keywords: Dexmedetomidine; Lignocaine; Upper Limb Orthopedic Surgery; Intravenous Regional Anaesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (Active Comparator): Patients will receive 3 mg/kg of 2% lignocaine (maximum dose 300 mg) alone diluted with normal saline 0.9% to make the final volume 30 ml
  Interventions: Drug: Lidocaine IV
- Group II (Active Comparator): Patients will receive 3 mg/kg of 2% lignocaine (maximum dose 300 mg) plus dexmedetomidine 0.25 μg/kg diluted with normal saline 0.9% to make the final volume 30 ml.
  Interventions: Drug: Dexmedetomidine Injectable Solution [Dexdomitor]; Drug: Lidocaine IV
- Group III (Active Comparator): Patients will receive 3 mg/kg of 2% lignocaine (maximum dose 300 mg) plus dexmedetomidine 0.5 μg/kg diluted with normal saline 0.9% to make the final volume 30 ml
  Interventions: Drug: Dexmedetomidine Injectable Solution [Dexdomitor]; Drug: Lidocaine IV

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Solution [Dexdomitor] — two different doses of dexemedetomidine (0.25 μg /kg and 0.5 μg/kg) as adjunct to lignocaine in intravenous regional anesthesia for upper limb orthopedic surgeries
  Arms: Group II; Group III
Drug: Lidocaine IV — Intravenous regional anaesthesia

SUMMARY:
A prospective randomized controlled double-blinded study will be conducted on 90 patients assigned randomly into three equal groups,

DETAILED DESCRIPTION:
After obtaining approval of the medical and ethical committee of Menoufia University & Nasser Institute for Research and Treatment, an informed and written consent from the patients, a prospective controlled randomized double blinded study will be performed

Sample size:

MedCalc® version 12.3.0.0 program "Ostend, Belgium" was used for calculations of sample size, statistical calculator based on 95% confidence interval and power of the study 80% with α error 5%, According to a previous study (13), showed that the duration of tourniquet time in group A was mean 51.60±5.157 and Group B was mean 53.80±4.773, with p-value >0.05, while Quality of block of excellent in group A 83.3% and group B 90%, it turns out that there is success in the group B compared to group A, but there is no difference. So it can be relied upon in this study, based on this assumption, sample size was calculated according to these values produced a minimal samples size of 86 cases were enough to find such a difference. Assuming a drop-out ratio of 5%, the sample size will be 90 cases, subdivided into three groups 30 cases in each group. Patients will be randomly categorized into three equal groups (30 patients each): The patients will be randomly allocated to one of these three groups, using a computer-generated sequence of random numbers and a sealed envelope technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA class I and II.
* Patients of either sex.
* Patients aged between 20-70 years.
* Patients scheduled for forearm and hand surgery lasting for about 60 minutes.

Exclusion Criteria:

* Patient with known hypersensitivity to any study medications.
* Patient with Severe peripheral vascular disease and neurological disease.
* Where use of tourniquet will be either not possible or contraindicated.
* Patient with Hemolytic diathesis specially sickle cell anemia, epilepsy, diabetes mellitus, hypertension, cardiovascular disease like myocardial infarction, cardiac arrhythmias, heart block and altered mentation.
* Procedures lasting for more than 90 min will be also not considered.
* Therapy with adrenergic receptor antagonist, calcium channel blocker and ACE inhibitors.
* Patient with impaired liver function.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
hollmen scale | 2 hours
  change from base line for the scale (scale from 1 to 4)
modified bromage scale | 2 hours
  change from baseline for the scale (scale from 0 to 4 )

SECONDARY OUTCOMES:
visual analogue score | 2 hours
  changes in the scale from 0 to 10
ramsey sedation score | 2 hours
  changes in the scale from 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Sadek AM Sadek, MD, Study Chair — Menoufia University
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No